CLINICAL TRIAL: NCT02515786
Title: Effects of Long-term Dry and Humidified Low-flow Oxygen Via Nasal Cannula on Nasal Mucociliary Clearance, Mucus Properties, Inflammation and Airway Symptoms in Patients
Brief Title: Effects of Long-term Dry and Humidified Low-flow Oxygen Via Nasal Cannula
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, Associate Professor of Physiotherapy, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 041/13
Record Dates: First submitted 2015-05-26; First posted 2015-08-05 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Respiratory Failure
Keywords: Chronic respiratory failure; Oxygen therapy; Nasal catheter; Mucociliary clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen humidification (Experimental): Oxygen by nasal catheter delivery will be humidified by bubles.
  Interventions: Other: oxygen humidification
- Dry oxygen (No Intervention): oxygen by nasal catheter delivery will be dry

INTERVENTIONS:
Other: oxygen humidification — humidification for oxygen delivered by nasal catheter
  Arms: oxygen humidification

SUMMARY:
During normal breathing, the upper and lower airways performs the priming of inspired gas: humidification, heating and filtering from nose to the bronchios for adequate gas exchange occurs in the lungs. Many patients with severe or advanced cardiopulmonary conditions (cystic fibrosis, chronic obstructive pulmonary disease, pulmonary hypertension, advanced heart failure among others) may develop chronic respiratory failure and require treatment with oxygen therapy. High fractions of inspired oxygen have been associated with deleterious effects on the nasal ciliary beating and nose mucociliary transport. At home assistance, the patient with chronic respiratory receives oxygen via nasal cannula to the patient has been applied with and without humidification, however, does not know the effects of these two types of dry and humidified administration on the mucosa of the nose, airways and lungs. The investigators will assess the subject in use of home oxygen therapy at baseline, 12 hours, 7 days 30 days, 12 months and 24 months.

DETAILED DESCRIPTION:
After agreeing to the terms of informed consent, the individual will be admitted to the study. The objective of this study was to evaluate the effects of humidified oxygen and not humidified nasal catheter (12-24 hours/day) on the nasal epithelium of patients with chronic respiratory failure by non-invasive tests in 36 volunteers, of both sexes aged ≥ 18 years with a medical indication for the use of home oxygen via nasal cannula on: (1) nasal mucociliary transport through the saccharin test, (2) the physical properties of nasal mucus by simulated cough machine and contact angle, (3) cellularity via nasal and total count differential white blood cell nasal lavage, (4) ph nasal lavage and exhaled breath condensate (5) quantification of cytokines in nasal lavage and (6) quality of life questionnaire with rhinosinusitis (SNOT20). Assessments will be performed at baseline, 12 hours, 7 days, 30 days, 12 months and 24 months of use. Volunteers will be recruited from three Basic Health Supervision of Cathedral Health, City Health Department, City of São Paulo.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged ≥ 18 years with a medical indication for the use of home low-flow oxygen via nasal cannula

Exclusion Criteria:

* inability to taste saccharin
* nasal surgery
* infection in the last 30 days (before the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
saccharin transit time test | First baseline measurement, 12 hours, 7 days, 30 days, 12 months and 24 months of use of home oxygen therapy
  The investigators evaluate the nasal MCC by measuring nasal saccharine transport time (STT). The subject is asked to avoid alcohol, tea and coffee for 6 hours and to eat or drink nothing for 2 hours before the measurements. The STT assessment is performed in a quiet room at a temperature of 21-22ºC and relative humidity of 63-71%. Subjects sat in a chair and are asked to maintain regular breathing, to avoid deep breathing, coughing, sneezing, sniffing or talking during STT measurements. Twenty-five µg saccharin particles are deposited 2 cm from the anterior end of the non-obstructed nostril and the timer is stopped at the first perception of sweet taste. The maximum delay between the deposition and perception is set at 60 minutes for non-detection.

OTHER OUTCOMES:
Analysis of Contact Angle of Mucus | First baseline measurement, 12 hours, 7 days, 30 days, 12 months and 24 months of use of home oxygen therapy
  In addition to the rheological properties of mucus, which imply on deformation and flow properties, and other characteristics as adhesiveness "wettabilidade" represents relevant physical properties in mucus transport by the cilia and cough . All biological fluid has the property of spreading when placed on a solid surface. As higher contact angle, lower is the "wettabilidade".
  Furthermore, the contact angle gives an inference adhesiveness, because the adhesion between the solid surface and specific mucus reflects the surface tension of the mucus and its contact angle. The contact angle is the angle formed between the tangent of the air-fluid interface and horizontal. The apparatus for measuring the contact angle is formed by a magnifying glass with hinged arm to move it laterally, forward and back. The magnifying glass has increased 25 times, with an eye that has a goniometer . The slide glass on which is deposited the
inflammation in the upper airway by analysis of nasal lavage | First baseline measurement, 12 hours, 7 days, 30 days, 12 months and 24 months. of use of home oxygen therapy
  Celularity and determination of IFN-α, IL-8, IL-10 and EGF (multiplex bead assay and ELISA) in nasal lavage. Celularity: the cell pellet is resuspended in one milliliter of phosphate buffer saline solution (PBS). Thereafter, 20 µl of the mixed solution is added to a Neubauer chamber, and the cells are counted using a 400x light microscope (Olympus CH2, Olympus America Inc., Palo Alto, USA). For differential cell counts, 100 µl of the mixed solution is centrifuged (96 g, 25°C, 6 min) to obtain a slide with two areas of cells that are stained with hematoxylin and eosin. Differential cell counts are performed with the aid of a 1000x light microscope (Olympus CH2, Olympus America Inc., Palo Alto, USA) by two different observers.
Upper airways symptoms by SNOT20 questionnaire | First baseline measurement, 12 hours, 7 days, 30 days, 12 months and 24 months of use of home oxygen therapy
  This is a questionnaire that aims to assess quality of life of patients with chronic upper airways symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Paulo HN Saldiva, Professor, Study Chair — School of Medicine University of Sao Paulo; Naomi K Nakagawa, Ph.D., Principal Investigator — School of Medicine University of Sao Paulo
Locations (1):
- School of Medicine University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Franchini ML, Athanazio R, Amato-Lourenco LF, Carreirao-Neto W, Saldiva PH, Lorenzi-Filho G, Rubin BK, Nakagawa NK. Oxygen With Cold Bubble Humidification Is No Better Than Dry Oxygen in Preventing Mucus Dehydration, Decreased Mucociliary Clearance, and Decline in Pulmonary Function. Chest. 2016 Aug;150(2):407-14. doi: 10.1016/j.chest.2016.03.035. Epub 2016 Apr 2. PMID 27048871